CLINICAL TRIAL: NCT06268236
Title: Electro-acupuncture to Treat Disorder of Consciousness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Fang Yuan, Principal Investigator, The Second Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BF2023-252
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Disorder of Consciousness; Electroacupuncture
Keywords: Acute brain injury; Disorder of consciousness; Electro-acupuncture; Awakening; Brain functional network
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-acupuncture group (Experimental): Patients in EA group receive acupuncture at Shuigou (also known as Renzhong, GV26) and Yintang (updated number GV24+, previous number GV29). Paired electrodes from the EA apparatus are clipped to the needle handles at Shuigou and Yintang. The electroacupuncture stimulation lasts for 30 minutes with a wave of rarefaction and condensation (10 Hz / 50 Hz) and a current intensity of the maximum withstand current within 7mA. All patients receive EA at 9 am for 30 minutes once a day for consecutive 14 days.
  Interventions: Other: Electroacupuncture
- Sham electro-acupuncture group (Sham Comparator): Patients in sham-EA group receive sham-EA at sham-Shuigou and sham-Yintang.Acupuncture needles are inserted into the adhesive pads but do not pierce the skin. Paired electrodes from the EA apparatus via sham connecting cords are clipped to the needle handles at sham-Shuigou and sham-Yintang. The sham connecting cords are similar in appearance to the normal ones, but the inner wires in sham connecting cords are cut off and cannot conduct electricity. All patients receive sham-EA at 9 am for 30 minutes once a day for consecutive 14 days.
  Interventions: Other: Sham electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — Electro-acupuncture at Shuigou and Yintang.
  Arms: Electro-acupuncture group
Other: Sham electroacupuncture — Sham-EA at sham-Shuigou and sham-Yintang.
  Arms: Sham electro-acupuncture group

SUMMARY:
With the rapid development of life support technology, more and more people can survive severe brain injury. Some survivors regain consciousness after a period of coma, however, many patients develop prolonged disorders of consciousness (DOC), which poses a therapeutic challenge for clinicians and a heavy burden for their families. The investigators design an Electro-acupuncture to treat disorder of consciousness (AcuDoc) trial with the aim of validating the clinical effect of electroacupuncture in treating DOC and exploring its therapeutic mechanisms by integrating EEG, neuroimaging, evoked potential tests, and behavioral assessments.

DETAILED DESCRIPTION:
The AcuDoc trial is a single-center, prospective, triple masking, randomized, sham electroacupuncture-controlled study. A total of 50 adult patients with DOC and 25 healthy subjects will be enrolled in the study . Patients will be randomized into electroacupuncture (EA) group or sham EA group (1:1). All patients will receive EA or sham-EA treatment in the supine position at 9 am for 30 minutes once a day for consecutive 14 days and healthy subjects will receive no treatments. The primary objective is to determine the therapeutic benefit of electroacupuncture on the recovery of consciousness in patients with DOC after a 2-week intervention. Key secondary objective is to investigate the effect of electroacupuncture on the circuitry of consciousness using a multimodal approach integrating EEG, neuroimaging (rs-fMRI, amide proton transfer imaging, intravoxel incoherent motion imaging, neurite orientation dispersion and density imaging), and evoked potentials (SEP, BAEP). Other secondary outcomes include the effect of EA on the assessment of brain-computer interface after a 2-week intervention and on the Glasgow Outcome Scale-Extended score at 30 days and 90 days .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. With cerebral damage due to TBI；
3. Diagnosed with UWS or MCS based on at least two CRS-R assessments;
4. From 4 to 16 weeks from the onset of brain injury;
5. Informed consent obtained.

Exclusion Criteria:

1. With a history of neurological or psychiatric disorder prior to the brain injury;
2. With uncontrolled seizures or status epilepticus;
3. Unstable vital signs and requiring the use of vasoactive agents;
4. With the use of general anesthetics or central acting sedative;
5. Without intact skin at acupoints or sham points;
6. Concomitant medical illness that would interfere with the outcome assessments and/or follow-up
7. Pregnant patients;
8. Currently participating in other investigational trials;
9. High likelihood of not adhering to the study treatment or the follow-up regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale - Revised score | after 14 days of EA or sham-EA treatment
  0 - 23, a higher score indicates a better level of consciousness

SECONDARY OUTCOMES:
phase locking value | after 14 days of EA or sham-EA treatment
  measured by electroencephalogram
amplitude of low-frequency fluctuation | after 14 days of EA or sham-EA treatment
  measured by resting-state functional magnetic resonance imaging
Amide proton transfer-weighted signal | after 14 days of EA or sham-EA treatment
  measured by amide proton transfer imaging
f value | after 14 days of EA or sham-EA treatment
  measured by intravoxel incoherent motion imaging
neurite density index | after 14 days of EA or sham-EA treatment
  measured by neurite orientation dispersion and density imaging
latency value of N20 | after 14 days of EA or sham-EA treatment
  measured by somatosensory evoked potential biomarkers
latency between III and V potentials | after 14 days of EA or sham-EA treatment
  measured by brainstem auditory evoked potential
Glasgow Outcome Scale-Extended score | 30 days after randomization
  1 - 8, a higher score indicates better functional recovery from brain injury
Glasgow Outcome Scale-Extended score | 90 days after randomization
  1 - 8, a higher score indicates better functional recovery from brain injury
brain-computer interface accuracy | after 14 days of EA or sham-EA treatment
  measured by electroencephalogram-based brain-computer interface experiment

CONTACTS AND LOCATIONS:
Overall Officials: Fang Yuan, PhD, Study Director — The Second Affiliated Hospital of Guangzhou University of Chinese Medicine
Locations (1):
- The Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The detailed datasets used and/or analyzed during the current study are available upon reasonable request.

REFERENCES:
- [Background] Thibaut A, Schiff N, Giacino J, Laureys S, Gosseries O. Therapeutic interventions in patients with prolonged disorders of consciousness. Lancet Neurol. 2019 Jun;18(6):600-614. doi: 10.1016/S1474-4422(19)30031-6. Epub 2019 Apr 16. PMID 31003899
- [Background] Laureys S, Celesia GG, Cohadon F, Lavrijsen J, Leon-Carrion J, Sannita WG, Sazbon L, Schmutzhard E, von Wild KR, Zeman A, Dolce G; European Task Force on Disorders of Consciousness. Unresponsive wakefulness syndrome: a new name for the vegetative state or apallic syndrome. BMC Med. 2010 Nov 1;8:68. doi: 10.1186/1741-7015-8-68. PMID 21040571
- [Background] Giacino JT, Ashwal S, Childs N, Cranford R, Jennett B, Katz DI, Kelly JP, Rosenberg JH, Whyte J, Zafonte RD, Zasler ND. The minimally conscious state: definition and diagnostic criteria. Neurology. 2002 Feb 12;58(3):349-53. doi: 10.1212/wnl.58.3.349. PMID 11839831
- [Background] Bruno MA, Vanhaudenhuyse A, Thibaut A, Moonen G, Laureys S. From unresponsive wakefulness to minimally conscious PLUS and functional locked-in syndromes: recent advances in our understanding of disorders of consciousness. J Neurol. 2011 Jul;258(7):1373-84. doi: 10.1007/s00415-011-6114-x. Epub 2011 Jun 16. PMID 21674197
- [Background] Steriade M, Nunez A, Amzica F. A novel slow (< 1 Hz) oscillation of neocortical neurons in vivo: depolarizing and hyperpolarizing components. J Neurosci. 1993 Aug;13(8):3252-65. doi: 10.1523/JNEUROSCI.13-08-03252.1993. PMID 8340806
- [Background] Timofeev I, Grenier F, Bazhenov M, Sejnowski TJ, Steriade M. Origin of slow cortical oscillations in deafferented cortical slabs. Cereb Cortex. 2000 Dec;10(12):1185-99. doi: 10.1093/cercor/10.12.1185. PMID 11073868
- [Background] Schiff ND. Recovery of consciousness after brain injury: a mesocircuit hypothesis. Trends Neurosci. 2010 Jan;33(1):1-9. doi: 10.1016/j.tins.2009.11.002. Epub 2009 Dec 1. PMID 19954851
- [Background] Giacino JT, Katz DI, Schiff ND, Whyte J, Ashman EJ, Ashwal S, Barbano R, Hammond FM, Laureys S, Ling GSF, Nakase-Richardson R, Seel RT, Yablon S, Getchius TSD, Gronseth GS, Armstrong MJ. Comprehensive systematic review update summary: Disorders of consciousness: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology; the American Congress of Rehabilitation Medicine; and the National Institute on Disability, Independent Living, and Rehabilitation Research. Neurology. 2018 Sep 4;91(10):461-470. doi: 10.1212/WNL.0000000000005928. Epub 2018 Aug 8. PMID 30089617
- [Background] Li H, Zhang X, Sun X, Dong L, Lu H, Yue S, Zhang H. Functional networks in prolonged disorders of consciousness. Front Neurosci. 2023 Feb 17;17:1113695. doi: 10.3389/fnins.2023.1113695. eCollection 2023. PMID 36875660
- [Background] Edlow BL, Claassen J, Schiff ND, Greer DM. Recovery from disorders of consciousness: mechanisms, prognosis and emerging therapies. Nat Rev Neurol. 2021 Mar;17(3):135-156. doi: 10.1038/s41582-020-00428-x. Epub 2020 Dec 14. PMID 33318675
- [Background] Rudolph M, Pelletier JG, Pare D, Destexhe A. Characterization of synaptic conductances and integrative properties during electrically induced EEG-activated states in neocortical neurons in vivo. J Neurophysiol. 2005 Oct;94(4):2805-21. doi: 10.1152/jn.01313.2004. Epub 2005 Jul 13. PMID 16014785
- [Background] Howell K, Grill E, Klein AM, Straube A, Bender A. Rehabilitation outcome of anoxic-ischaemic encephalopathy survivors with prolonged disorders of consciousness. Resuscitation. 2013 Oct;84(10):1409-15. doi: 10.1016/j.resuscitation.2013.05.015. Epub 2013 Jun 6. PMID 23747956
- [Background] Perez P, Valente M, Hermann B, Sitt J, Faugeras F, Demeret S, Rohaut B, Naccache L. Auditory Event-Related "Global Effect" Predicts Recovery of Overt Consciousness. Front Neurol. 2021 Jan 8;11:588233. doi: 10.3389/fneur.2020.588233. eCollection 2020. PMID 33488494
- [Background] Threlkeld ZD, Bodien YG, Rosenthal ES, Giacino JT, Nieto-Castanon A, Wu O, Whitfield-Gabrieli S, Edlow BL. Functional networks reemerge during recovery of consciousness after acute severe traumatic brain injury. Cortex. 2018 Sep;106:299-308. doi: 10.1016/j.cortex.2018.05.004. Epub 2018 May 12. PMID 29871771
- [Background] Demertzi A, Tagliazucchi E, Dehaene S, Deco G, Barttfeld P, Raimondo F, Martial C, Fernandez-Espejo D, Rohaut B, Voss HU, Schiff ND, Owen AM, Laureys S, Naccache L, Sitt JD. Human consciousness is supported by dynamic complex patterns of brain signal coordination. Sci Adv. 2019 Feb 6;5(2):eaat7603. doi: 10.1126/sciadv.aat7603. eCollection 2019 Feb. PMID 30775433